CLINICAL TRIAL: NCT00843219
Title: Motion Correction of Positron Emission Tomography (PET) Data Using Amplitude Gating
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: 2008-0851
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2012-01

CONDITIONS: Lung Cancer
Keywords: Lung; Lung Cancer; Non-small cell Lung Cancer; NSCLC; Motion Correction; PET/CT Scan; PET; Positron Emission Tomography; CT; Computed Tomography; Amplitude Gating
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PET/CT Scan
  Interventions: Procedure: PET/CT Scan

INTERVENTIONS:
Procedure: PET/CT Scan — PET/CT scan performed with elastic belt around lower chest/upper abdomen to track breathing motion.
  Other Names: Positron Emission Tomography; Positron Emission Tomography/Computed Tomography; Computed Tomography

SUMMARY:
Objectives:

Evaluation of an amplitude based gated Positron Emission Tomography (PET) data acquisition system for all GE Discovery Positron Emission Tomography/ Computed Tomography (PET/CT) scanners.

DETAILED DESCRIPTION:
Routine PET/CT scans are taken while patients are breathing normally. The motions made by breathing can reduce the image quality of the scan. Minimizing the effects of this motion by taking the images and processing the scans differently may improve the image quality.

The PET/CT Scan:

If you agree to take part in this study, an elastic belt will be placed around your lower chest/upper abdomen before your routine PET/CT scan. This belt is used to track your breathing motion. This information will be used to help process the scan.

Your PET/CT scan will be performed as usual. During the scan, researchers will focus on your lower chest/upper abdomen (areas that experience breathing motion). Having to focus on this area might extend the scan by up to 10 minutes.

The additional scan time will not increase your radiation exposure since only PET scanning will be performed.

Length of Study:

Your participation on this study will be complete when your scheduled PET/CT scan is complete.

This is an investigational study. The imaging focused on your lower chest/upper abdomen during the scan is investigational.

Up to 26 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with lung or liver lesions measuring 0.5-2cm in diameter will be considered.
2. Patients that are scheduled to be imaged in the PET/CT suite at the Mays Building will only be considered.

Exclusion Criteria:

1. Pediatric patients (younger than 18 years) will be excluded.
2. Patients that cannot tolerate being scanned for an additional 10 minutes with arms above their head will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals over the age of 18 with non-small cell lung cancer (NSCLC) and are scheduled to have a positron emission tomography/computed tomography (PET/CT) scan.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2009-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Mean Difference Between Gated + Ungated PET/CT Scans | Scheduled PET/CT scans extended by 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Osama R Mawlawi, PHD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org